CLINICAL TRIAL: NCT01339884
Title: An Open Label Clinical Pilot Study of Resveratrol as Treatment for Friedreich Ataxia
Brief Title: A Study of Resveratrol as Treatment for Friedreich Ataxia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Friedreich's Ataxia Research Alliance (Other)
Responsible Party: Principal Investigator, Martin Delatycki, Prof Martin Delatycki, Murdoch Childrens Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10358B
Record Dates: First submitted 2011-04-14; First posted 2011-04-21 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Friedreich Ataxia
Keywords: Friedreich ataxia; Resveratrol; Frataxin; Cardiomyopathy; Oxidative stress
MeSH Terms: conditions — Friedreich Ataxia; Cardiomyopathies | interventions — Resveratrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resveratrol, 1g daily (Active Comparator): 15 participants will receive resveratrol 1g daily
  Interventions: Drug: Resveratrol
- Resveratrol, 5g daily (Active Comparator): 15 participants will receive resveratrol, 5g daily
  Interventions: Drug: Resveratrol

INTERVENTIONS:
Drug: Resveratrol — Resveratrol 1g daily (500mg twice daily) for 12 weeks Resveratrol 5 daily (2.5g twice daily) for 12 weeks

SUMMARY:
The purpose of this study is to determine the effect of two doses of resveratrol taken for a 12 week period, on frataxin levels in individuals with Friedreich ataxia. This study will also measure the effect of resveratrol on markers of oxidative stress, clinical measures of ataxia, and cardiac parameters.

DETAILED DESCRIPTION:
Resveratrol shows promise as an agent for the treatment of Friedreich ataxia due to its antioxidant properties, neuroprotective effects, and ability to increase frataxin levels in vitro and in vivo. This clinical pilot study aims to determine the effect of two doses of resveratrol (1g/day and 5g/day) taken for 12 weeks, on frataxin levels in individuals with Friedreich ataxia. Additional outcome measures include the effect of resveratrol on markers of oxidative stress, clinical measures of ataxia , and cardiac parameters (including relative wall thickness and left ventricular mass index).

ELIGIBILITY:
Inclusion Criteria:

* Adults with Friedreich ataxia due to homozygosity for the GAA repeat expansion in intron 1 of the FXN gene
* Functional stage on the Ataxia subscale of the FARS of 1 or higher

Exclusion Criteria:

* Women who are pregnant or lactating
* Active arrythmias or significant cardiac insufficiency
* Use of idebenone, Coenzyme Q or vitamin E within 30 days prior to enrolment
* Use of amiodarone or other medications which may have clinically significant drug interactions that cannot be safely monitored

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Lymphocyte frataxin level | 12 weeks
  Change in lymphocyte frataxin levels at 12 weeks compared to baseline

SECONDARY OUTCOMES:
Oxidative stress markers | 12 weeks
  Oxidative stress, as measured by a) plasma F2-isoprostanes and b) urinary 8-hydroxyl-2-deoxyguanosine levels at 12 weeks compared to baseline
Clinical rating scales of ataxia | 12 weeks
  Clinical rating scales of ataxia at 12 weeks will be compared to baseline. This will include: a) Friedreich Ataxia Rating Scale (FARS) b) International Cooperative Ataxia Rating Scale (ICARS) c) Scale for the Assessment and Rating of Ataxia (SARA) d) Friedreich Ataxia Functional Composite
Echocardiogram measures | 12 weeks
  Changes in structural and functional 3D echocardiogram measures from baseline to 12 weeks will be reported
Pharmacokinetic studies of resveratrol | First 2 hours post dose
  Pharmacokinetic data will be collected 45, 90 and 120 minutes after the first dose of resveratrol. Plasma concentration of resveratrol and its sulfate and glucuronide metabolites will be measured in ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Delatycki, MBBS PhD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Monash Medical Centre, Southern Health, Clayton, Melbourne, Victoria, Australia